CLINICAL TRIAL: NCT01445340
Title: Phase I Study of Topical Romidepsin (Depsipeptide) in Early Stage Cutaneous T-Cell Lymphoma
Brief Title: Topical Romidepsin to Treat Early-Stage Cutaneous T-Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070133; 07-C-0133; NCT00477698 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-06-29

CONDITIONS: Mycosis Fungoides; Cutaneous T-Cell Lymphoma; Neoplasms
Keywords: Topical Depsi; Cutaneous T Cell Lymphoma; CTCL; Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Neoplasms | interventions — romidepsin

INTERVENTIONS:
Drug: Romidepsin (FR901228)

SUMMARY:
Background:

* Cutaneous T-cell lymphoma (CTCL) is a rare, slow-growing form of skin cancer. The cancer cells are found in red, scaly patches that may sometimes itch.
* Early-stage CTCL is usually treated with topical therapies, which may lose effectiveness over time and have adverse effects, such as risk of secondary skin cancers and difficulty of use.
* Romidepsin is an experimental drug that, given through a vein, has improved CTCL in some patients with later stages of the disease.
* A topical ointment form of romidepsin may be helpful in treating early-stage CTCL.

Objectives:

* To determine the highest tolerated dose of topical romidepsin that can be given to patients with early-stage CTCL.
* To evaluate the effectiveness of topical romidepsin in patients with early-stage CTCL.
* To determine how the body handles topical romidepsin.

Eligibility:

-Patients 18 of age and older with early-stage CTCL.

Design:

* Study Part 1: Successive groups of 3 patients are treated with increasingly higher concentrations of topical romidepsin until the highest tolerated dose is found.
* Study Part II: The highest tolerated dose, as determined in Part I, is applied to larger areas of skin in another group of patients.
* All study participants apply the study medicine to their skin three times a day for 4 weeks.
* During treatment, participants are monitored at weeks 2 and 4 with a history and physical examination, blood tests, electrocardiogram, skin biopsies and photographs of the skin.
* After stopping treatment, participants return to the clinic at weeks 6 and 8 for blood tests and to see how the study medication is affecting the body.

DETAILED DESCRIPTION:
Background:

* Romidepsin is a histone deacetylase inhibitor which has demonstrated efficacy and tolerability as an infusion in later stages of cutaneous T-cell lymphoma (CTCL).
* Early stages of CTCL are typically treated with skin-directed therapies, which may lose efficacy over time and have adverse effects (i.e. risk of secondary skin cancers, difficulty of use).
* A topical form of romidepsin may be helpful in the treatment of early-stage CTCL.

Objectives:

* Primary - To define the maximal tolerated dose (MTD) of topical romidepsin for early-stage CTCL when administered three times weekly, then escalated first in concentration, followed by increased frequency and lastly over increasing body surface areas.
* Secondary - To assess histone acetylation in topical romidepsin-treated skin.
* Secondary - To assess in a pilot fashion clinical efficacy of topical romidepsin in early stage cutaneous T-cell lymphoma.
* Secondary - To perform pharmacokinetic monitoring of blood levels of romidepsin in topically treated patients.

Eligibility:

-Patients age greater than or equal to 18 with confirmed early-stage (stage IA, IB, or IIA) cutaneous T-cell lymphoma.

Design:

* A Cohorts of Three design to define the MTD of topical romidepsin in Aquaphor ointment initially applied overnight, three times weekly for 4 weeks, then escalated first in concentration, followed by increased frequency and lastly over increasing body surface areas.
* Skin toxicities, systemic toxicities, and disease response will be assessed throughout the study.
* The primary focus of the first part of the protocol will be to evaluate local skin toxicity, beginning with dose level 1 of 0.05 percent topical romidepsin on 25 cm(2) target area (0.005 mg/ cm(2). If tolerated, progress to higher dose levels of 0.25 percent (0.025 mg/ cm(2); dose level 2) and then 0.5 percent (0.05 mg/ cm(2); dose level 3) topical romidepsin on 25 cm(2) target area. Systemic toxicity will also be monitored.
* To date, we have completed the first 4 dose levels and have not yet established cutaneous MTD. To achieve this, we will proceed to the second part of the protocol, which will increase the concentration to 1%, then increase the frequency to daily application, then progress to 2% concentration, then 4% concentration, and then applying to progressively larger body surface areas. Our aim is to more fully address systemic toxicity by increasing drug concentration, application frequency, and body surface area (BSA) treated. We will utilize topical romidepsin at the MTD on increasing BSA (lesional & nonlesional skin): multiple lesions up to 3% BSA (dose level 4), multiple lesions up to 25% BSA (dose level 7A), 50% BSA (dose level 7B), and 75% or > BSA (dose level 7C).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have a pathologically confirmed diagnosis of CTCL based on a skin biopsy, utilizing standard histological criteria based on cytological, architectural, and immunophenotypic findings. In cases with equivocal histological features, the diagnosis may be verified or confirmed through the use of clonal T-cell gamma gene rearrangement, as detected by PCR amplification and primer sets specific for the T-cell receptor gamma chain genes.
  2. Patients must have early stage CTCL (Stage IA, IB, or IIA as defined by TNM staging system).
  3. Patients must:

     1. be age greater than or equal to 18 years.
     2. have evaluable disease.
     3. have a performance status of ECOG 0-1.
     4. be either on no therapy or only on topical therapy for early stage CTCL. Patients must have stopped light therapy (i.e. PUVA, UVB) for at least 2 weeks prior to the use of study medication. Patients must have stopped topical therapies (i.e. corticosteroids or nitrogen mustard) to designated target sites or areas to be treated with study medication for at least 2 weeks prior to the use of study medication. (Topical therapies for CTCL may be continued to non-adjacent, non-target lesions while on protocol.) Patients may have received other HDACI therapy but must have stopped systemic therapy 4 weeks prior to use of study medication.
     5. be able to give written informed consent.
     6. be willing to return to the National Cancer Institute for follow-up.
  4. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. The effects of romidepsin on the developing human fetus are unknown. For this reason and because HDAC Inhibitor agents are known to be teratogenic, patients that are pregnant or lactating will be excluded from this trial.
  5. Laboratory values:

     Within 7 days prior to registration: absolute neutrophil count greater than or equal to 1000/microL, platelets greater than or equal to 100,000/microL, bilirubin (total and direct) less than or equal to 1.5 times upper limit of normal, and AST less than or equal to 3 times upper limit of normal, creatinine less than or equal to 1.5 times upper limit of normal, or documented creatinine clearance of greater than or equal to 60mL/min
  6. Cardiac findings:

Within 4 weeks of registration: ECG [patients should not have QTc prolongation (greater than 480 msec) and/or rhythm abnormality; allowance of other EKG changes will be at discretion of the investigator based on consultation with a cardiologist] and echocardiogram [demonstrating normal ejection fraction].

EXCLUSION CRITERIA:

1. Prior or concurrent malignancies that have not been curatively treated with the exception of malignancies that have been curatively treated and without recurrence in the preceding 5 years, non-melanoma skin cancers, low grade cervical cancer and prostate cancer.
2. Current or previous CNS metastasis.
3. Chemotherapy within 4 weeks, 6 weeks for nitrosoureas or mitomycin C, and 8 weeks for UCN-01.
4. HIV seropositivity.
5. Pregnant or breast-feeding patients.
6. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Use of known CYP3A4 inhibitors within 3 days prior to receiving romidepsin ointment treatment.

Inclusion of Women and Minorities:

Subjects from both genders and all racial/ethnic groups are eligible for this study if they meet the eligibility criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-04-21; Study Completion 2012-06-29 (Actual)

PRIMARY OUTCOMES:
To define the maximal tolerated dose of topical romidepsin.

SECONDARY OUTCOMES:
To assess histone acetylation in topical romidepsin-treated skin, to assess in a pilot fashion clinical efficacy of topical romidepsin in early stage CTCL and to perform pharmacokinetic monitoring of blood levels of topical romidepsin.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi H Kong, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ueda H, Nakajima H, Hori Y, Goto T, Okuhara M. Action of FR901228, a novel antitumor bicyclic depsipeptide produced by Chromobacterium violaceum no. 968, on Ha-ras transformed NIH3T3 cells. Biosci Biotechnol Biochem. 1994 Sep;58(9):1579-83. doi: 10.1271/bbb.58.1579. PMID 7765477
- [Background] Kitazono M, Chuman Y, Aikou T, Fojo T. Construction of gene therapy vectors targeting thyroid cells: enhancement of activity and specificity with histone deacetylase inhibitors and agents modulating the cyclic adenosine 3',5'-monophosphate pathway and demonstration of activity in follicular and anaplastic thyroid carcinoma cells. J Clin Endocrinol Metab. 2001 Feb;86(2):834-40. doi: 10.1210/jcem.86.2.7196. PMID 11158054
- [Background] Ueda H, Manda T, Matsumoto S, Mukumoto S, Nishigaki F, Kawamura I, Shimomura K. FR901228, a novel antitumor bicyclic depsipeptide produced by Chromobacterium violaceum No. 968. III. Antitumor activities on experimental tumors in mice. J Antibiot (Tokyo). 1994 Mar;47(3):315-23. doi: 10.7164/antibiotics.47.315. PMID 8175484